CLINICAL TRIAL: NCT03484403
Title: Benefit of Lumbar Bracing for Chronic Low Back Pain Due to Degenerative Disc Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dallas VA Medical Center (U.S. Federal Agency)
Collaborators: Aspen Medical Products (Other)
Responsible Party: Principal Investigator, Thiru Annaswamy, Professor, PM&R, Principal Investigator, Staff Physician, Dallas VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-088
Record Dates: First submitted 2018-03-23; First posted 2018-03-30 (Actual); Results first posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2023-04

CONDITIONS: Degenerative Disc Disease; Lumbar Spondylosis; Low Back Pain
MeSH Terms: conditions — Intervertebral Disc Degeneration; Spondylosis; Low Back Pain

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized controlled trial. Blinding of the subjects is not possible because a back brace is a visibly obvious intervention. In addition, since we are evaluating the adherence of back brace wear, blinding of the investigator is also not possible. Therefore, this study will be an unblinded RCT.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Study participants will not receive a back brace but will receive back school education and the same physical therapy exercise instruction as the treatment group.
  Interventions: Behavioral: Back school
- Treatment Group (Experimental): Study participants in this group will receive a lumbar support back brace and will receive back school education and the same physical therapy exercise instruction as the control group.
  Interventions: Other: Lumbar back brace; Behavioral: Back school

INTERVENTIONS:
Other: Lumbar back brace — A brace that supports the lumbar region of the spine.
  Arms: Treatment Group
Behavioral: Back school — Back school consists of patient education physical therapy exercise instruction.

SUMMARY:
The main objectives of this study are to evaluate the benefits of back bracing in the symptomatic management of patients with CLBP due to degenerative lumbar disc disease. The plan is to study patients with uncomplicated CLBP without symptoms of radiculopathy or neurogenic claudication.

The secondary objectives of the study are to evaluate if a back brace provides any additive benefit to usual care consisting of exercise and patient education in patients with CLBP due to degenerative disc disease.

Specific Aim 1. To evaluate the effectiveness of back brace to improve pain and patient-reported functional measures in patients with uncomplicated CLBP due to degenerative disc and degenerative joint disease without associated symptoms of neurogenic claudication or lumbosacral radiculopathy.

Hypothesis 1. Back brace in addition to usual care will provide statistically significant improvement in pain and functional measures compared to usual care alone.

Specific Aim 2. To evaluate the adherence to back brace wear instructions in patients with uncomplicated CLBP due to degenerative disc and degenerative joint disease without associated symptoms of neurogenic claudication or lumbosacral radiculopathy Hypothesis 2. Patients with CLBP, due to degenerative disc and degenerative joint disease without associated symptoms of neurogenic claudication or lumbosacral radiculopathy, who are prescribed a back brace, will demonstrate clinically acceptable rates of adherence to brace wear instructions.

DETAILED DESCRIPTION:
Physiatrists use back braces (lumbar support, back corset, semi-rigid brace, and lumbar orthotic) for symptomatic management of patients' chronic low back pain (CLBP) despite very poor evidence supporting their use in the few published studies that have examined them. Evidence supporting back braces in other populations, such as pregnant women, and patients with sub-acute or acute low back pain, is better established. However, the benefits of back braces in the CLBP population are very unclear.

A Cochrane review on the role of lumbar supports in treating chronic LBP revealed that limited evidence was available, which led to the conclusion that, "it remains unclear whether lumbar supports are more effective than no or other interventions for treating low-back pain." The research emphasized the need for high quality randomized trials evaluating the effectiveness of back braces, and also recommended that compliance of brace wear be monitored.

The mechanism by which back braces might help patients with CLBP is also unclear. The semi-rigid design of the commonly used back brace does not mechanically limit movement enough to suggest that movement limitation is the mechanism by which back braces provide relief. However, some studies have suggested that back braces help patients with CLBP by providing postural support or a kinesthetic reminder of their posture. Using posturography, Munoz et al., studied the forces applied by lumbar bracing and concluded that back braces seem to help by improving the quality of balance strategy used by the patient. Another mechanism by which back braces are believed to help patients is by providing warmth underneath the brace.

There is poor published information regarding adherence to instructions (compliance) about the use of back braces. Based on the investigators' anecdotal clinical experience, adherence rates vary widely among patients who are prescribed back braces, ranging from non-use to constant use around the clock. Poor adherence to instructions can be a significant factor resulting in inconclusive evidence supporting the role of back brace in patients with CLBP. A recent study showed that a strong predictor for consistent adherence to back brace usage was a positive attitude towards it. In this study, positive attitude towards the back brace explained 41% of the variance in outcomes. In addition, investigators found that perceived benefit from the brace outweighed any subjective discomfort.

Back braces have been used as adjunctive therapy in addition to other conservative care options. A recent study evaluated the cumulative effect of bracing to exercise and found that bracing helps to increase trunk stiffness and augments muscle contractions, which may remind the patients to better comply with exercise instructions. This suggested a potential synergistic effect of bracing and exercise in the management of patients with CLBP.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of lumbar degenerative disc disease or joint disease
* Low back pain > 6 weeks
* Uncomplicated low back pain without symptoms of pain radiating below the knee

Exclusion Criteria:

* Lumbar radiculopathy
* Neurogenic claudication
* Spondylolisthesis with instability
* Previous lumbar spine surgery
* Recent (<1 year) brace use or physical therapy program
* No active psychiatric illness

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2015-12-14 (Actual); Primary Completion 2019-09-10 (Actual); Study Completion 2019-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thiru Annaswamy, M.D., Principal Investigator — Dallas VA Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] O'Keeffe M, Nolan D, O'Sullivan P, Dankaerts W, Fersum K, O'Sullivan K. Re: Aleksiev AR. Ten-year follow-up of strengthening versus flexibility exercises with or without abdominal bracing in recurrent low back pain. Spine (Phila Pa 1976). 2014 Nov 15;39(24):E1495-7. doi: 10.1097/BRS.0000000000000620. No abstract available. PMID 25387146
- [Background] Roelofs PD, Bierma-Zeinstra SM, van Poppel MN, van Mechelen W, Koes BW, van Tulder MW. Cost-effectiveness of lumbar supports for home care workers with recurrent low back pain: an economic evaluation alongside a randomized-controlled trial. Spine (Phila Pa 1976). 2010 Dec 15;35(26):E1619-26. doi: 10.1097/BRS.0b013e3181cf7244. PMID 20823783
- [Background] Munoz F, Salmochi JF, Faouen P, Rougier P. Low back pain sufferers: is standing postural balance facilitated by a lordotic lumbar brace? Orthop Traumatol Surg Res. 2010 Jun;96(4):362-6. doi: 10.1016/j.otsr.2010.01.003. Epub 2010 May 7. PMID 20452305
- [Background] van Duijvenbode IC, Jellema P, van Poppel MN, van Tulder MW. Lumbar supports for prevention and treatment of low back pain. Cochrane Database Syst Rev. 2008 Apr 16;2008(2):CD001823. doi: 10.1002/14651858.CD001823.pub3. PMID 18425875
- [Background] Pennick V, Liddle SD. Interventions for preventing and treating pelvic and back pain in pregnancy. Cochrane Database Syst Rev. 2013 Aug 1;(8):CD001139. doi: 10.1002/14651858.CD001139.pub3. PMID 23904227
- [Background] Calmels P, Queneau P, Hamonet C, Le Pen C, Maurel F, Lerouvreur C, Thoumie P. Effectiveness of a lumbar belt in subacute low back pain: an open, multicentric, and randomized clinical study. Spine (Phila Pa 1976). 2009 Feb 1;34(3):215-20. doi: 10.1097/BRS.0b013e31819577dc. PMID 19179915
- [Background] Podichetty VK, Varley ES. Re: Oleske D M, Lavender S A, Andersson G B, et al. Are back supports plus education more effective than education alone in promoting recovery from low back pain? Results from a randomized clinical trial. Spine 2007;32:2050-7. Spine (Phila Pa 1976). 2008 Feb 1;33(3):349-50. doi: 10.1097/BRS.0b013e31816244db. No abstract available. PMID 18303469
- [Derived] Annaswamy TM, Cunniff KJ, Kroll M, Yap L, Hasley M, Lin CK, Petrasic J. Lumbar Bracing for Chronic Low Back Pain: A Randomized Controlled Trial. Am J Phys Med Rehabil. 2021 Aug 1;100(8):742-749. doi: 10.1097/PHM.0000000000001743. PMID 33789322

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with a diagnosis of lumbar degenerative disc disease or joint disease were recruited from the Physical Medicine and Rehabilitation clinic at the Veterans Affairs Medical Center, and were included in the study if they met the study criteria.
Pre-assignment Details: 2 participants withdrew after enrollment
Period: Overall Study
Arm/Group | Control Group | Treatment Group
Started | 34 | 25
Completed | 28 | 21
Not Completed | 6 | 4
Not completed — Withdrawal by Subject | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Treatment Group | Total
Number analyzed (Participants) | 34 | 25 | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 21 | 51
  >=65 years | 4 | 4 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.5 (13.1) | 47.6 (15.1) | 48.9 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 3 | 11
  Male | 26 | 22 | 48
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/Black | 17 | 16 | 33
  Caucasian/White | 12 | 8 | 20
  Hispanic or Latino | 5 | 1 | 6
Region of Enrollment [Number; unit: participants]
  United States | 34 | 25 | 59
Pain Disability Questionnaire [Mean (Standard Deviation); unit: units on a scale] — The Pain Disability Questionnaire (PDQ) allows patients to rate their ability to complete specific tasks on a 10-cm visual analog scale (15 questions) ranging from having no problems with the task (zero) to being unable to complete it at all (ten).
  Psychosocial and functional component subscores and the total score are calculated based on the responses. The maximum total score is 150; the maximum psychosocial subscore is 60; and the maximum functional subscore is 90. Lower scores indicate less pain-related disability.
  units on a scale | 79.26 (23.29) | 80.65 (23.33) | 79.96 (23.31)

OUTCOME MEASURES:

1. Primary Outcome: Pain Diary
Description: Patients rate their weekly pain on a scale from 0-10. Lower values indicate better outcomes.
  Average weekly pain scores were compared from baseline to 6 week mark.
Time Frame: Change between baseline and each week for 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 34 | 25
units on a scale | 6.71 (1.56) | 5 (1.78)

2. Primary Outcome: Pain Disability Questionnaire
Description: Measures how pain affects the patients lifestyle and participation in activities.
  Ranges from 0-150. Higher values indicate worse outcome.
Time Frame: These assessments were made at baseline (T₀), 6 wks (T₁), 12 wks (T₂), and 6 mos (T₃). Change between baseline and each follow-up visit (6 weeks, 12 weeks and 6 months).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 34 | 25
units on a scale
  Baseline | 79.26 (23.29) | 80.65 (23.33)
  6-weeks | 73 (24) | 78.2 (24)
  12-weeks | 68 (24) | 79.2 (25)
  6-months | 59.6 (25) | 80 (25.1)

3. Primary Outcome: PROMIS Instrument Questionnaire
Description: Patient reported outcome measure that measures how their pain problem is interfering with their quality of life and function. Higher scores indicate worse outcomes. Higher scores = more pain interference with function, range = 0-112
Time Frame: Change between baseline and each follow-up visit (6 weeks, 12 weeks and 6 months)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 34 | 25
units on a scale
  Baseline | 53.82 (20.74) | 52.7 (18.37)
  6-weeks | 49 (21) | 53 (19)
  12-weeks | 47 (21.2) | 56 (22)
  6-months | 42.2 (22.2) | 61.9 (24)

4. Primary Outcome: European Qualify of Life (EQ-5D) Questionnaire
Description: Measures quality of life for pre- and post comparisons. Higher scores indicate better outcomes. higher scores = poorer quality of life, range = 0-10
Time Frame: Change between baseline and each follow-up visit (6 weeks, 12 weeks and 6 months)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 34 | 25
units on a scale
  Baseline | 3.82 (1.6) | 4.13 (1.75)
  6-weeks | 3.6 (1.5) | 4.3 (1.8)
  12-weeks | 3.4 (1.7) | 4.8 (1.9)
  6-months | 3 (1.5) | 5 (2.2)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected till the final time point of the study (6 months from baseline visit)
Arm/Group | Control Group | Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/25
Other Adverse Events (participants affected / at risk) | 0/34 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-01-02): https://cdn.clinicaltrials.gov/large-docs/03/NCT03484403/Prot_SAP_000.pdf
  • Informed Consent Form (2018-11-09): https://cdn.clinicaltrials.gov/large-docs/03/NCT03484403/ICF_001.pdf